CLINICAL TRIAL: NCT04148924
Title: Comparison Between the Assessment of Anxious and Depressive Symptomology by the Patient and the Evaluation of the Patient's Symptoms by Caregivers: a Pilot Study Carried Out in a French Palliative Care Unit.
Brief Title: Comparison Between the Assessment of Anxious and Depressive Symptomology
Acronym: EDAPAL
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL19_0301
Record Dates: First submitted 2019-10-31; First posted 2019-11-04 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: End Stage Disease
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Patients: Anyone who is hospitalized in the palliative care service of the Lyon Sud Hospital Center.
  Interventions: Other: Questionnaire
- Doctors: Doctors taking care of patients in the study will be solicited by the research nurse or a study investigator.
  Interventions: Other: Medical staff questionnaire
- Nurses: Nurses taking care of patients in the study will be solicited by the research nurse or a study investigator.
  Interventions: Other: Medical staff questionnaire
- Caregivers: Caregivers taking care of patients in the study will be solicited by the research nurse or a study investigator.
  Interventions: Other: Medical staff questionnaire

INTERVENTIONS:
Other: Questionnaire — Patients complete a questionnaire for assess their symptoms like anxiety and depression.
  These questionnaires contains:
  * socio-demographic characteristics : sex, age, type and stage of cancer, performans status
  * ESAS : Edmonton Symptom Assessement Scale is a validated tool for assessment of several symptoms
  * HADS - A : Hospital Anxiety and Depression scale includes 2 subscales which assess anxiety (HADS-A) and depression (HADS-D)
  * BEDS : Brief Edimburg depression Scale is s a relevant scale for assess depression in palliative care patients.
  * Questions on the assessment, the treatment and difficulties in management of anxious and depressive symptoms.
  The evaluation will be realized in the first days of hospitalization (72 hours).
  Groups: Patients
Other: Medical staff questionnaire — Questionnaire is different from caregivers. The evaluation will be realized in the first days of hospitalization (72 hours).
  Physicians, nurses and caregivers complete another questionnaire. The physician questioned will be the doctor of unit having received the patient, or the doctor of the mobile team of palliative care having admitted the patient in the unit.
  These questionnaires contains:
  * socio-demographic characteristics : sex, age, type and stage of cancer, performans status
  * ESAS : Edmonton Symptom Assessement Scale is a validated tool for assessment of several symptoms
  Groups: Caregivers; Doctors; Nurses

SUMMARY:
In palliative care, anxiety and depression in advanced cancer are under evaluated, under diagnosed and therefore under treated. 5 to 30% of patients present anxious and depressive disorders.

Physical symptoms are easy to assess. But in palliative care it is important to take care of moral suffering.

However, evaluation and management of patient's anxiety and depressive symptoms are difficult for physicians and caregivers.

The investigators would like to specifically compare the patient's evaluation of anxious and depressive symptomatology in palliative care with the evaluation by the physician, the nurse and the caregiver.

Then the investigators will try to collect the caregivers's difficulties in the management of anxious and depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

Patients :

* Adult patients (18 years and over)
* Advanced cancer stage
* Patients hospitalized less than 72 hours in Lyon Sud palliative care unit
* Sufficient general conditions to complete survey
* Absence of cognitive disorders
* Agreement to participate at the study

Medical Staff:

- Working full time or part time in the USP or the PMSC of CHLS

Exclusion Criteria:

Patients :

* Minor patients
* Patients hospitalized more than 72 hours in Lyon Sud palliative care unit
* Presence of cognitive disorders
* Alteration of general conditions
* Refusal to participate at the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All patients hospitalized in our palliative care unit
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-11-15 (Actual); Primary Completion 2020-11-13 (Actual); Study Completion 2020-11-13 (Actual)

PRIMARY OUTCOMES:
Comparison of the anxious and depressive symptomatology of hospitalized patients in palliative care unit (USP) evaluated on the one hand by the patient himself and on the other hand, in hetero evaluation, by caregivers. | 72 hours
  The Edmonton Symptom Assessment Scale (ESAS) will be used for assess anxiety and depression intensity. The ESAS is a self-reported outcome tool assessing the intensity of nine symptoms (pain, tiredness, nausea, depressive mood, anxiety, drowsiness, lack of appetite, wellbeing, and breathlessness). Intensity is rated using 10-point Likert-scales from "no-symptom" (scored 0) to "worst possible symptom" (scored 10)
  The difference of evaluation for anxiety and depressive symptoms is considere significant when there are two points and more between ESAS patient's and ESAS caregivers'.

CONTACTS AND LOCATIONS:
Overall Officials: Audrey FAWOUBO, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Lyon Sud, Pierre-Bénite, France